CLINICAL TRIAL: NCT01787045
Title: Effect of Early Physical Activity on Skeletal Muscle Signaling Pathways Controlling Protein Turnover in Patients With Sepsis.
Brief Title: Early Physical Therapy in Patients With Sepsis
Acronym: EARTH-ICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EarlyPTProtocol1
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: SEPTIC SHOCK; SEPSIS SYNDROME; Multiple Organ Dysfunction Syndrome
Keywords: SEPSIS
MeSH Terms: conditions — Shock, Septic; Systemic Inflammatory Response Syndrome; Multiple Organ Failure; Sepsis | interventions — Early Ambulation; Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Early and Active Physical Therapy will be performed by physiotherapist twice a day. During first week patients will be positioned in chair or bed and performed cycle-ergometer exercise during 30 min.
  Our physiotherapy protocol will be continued until Intensive Care Unit (ICU) discharge.
  Interventions: Other: Early and Active Physical Therapy; Other: Passive Range of Motion
- Control Group (Other): Routinary Passive Range of Motion will be performed by physiotherapist 20 min and twice a day until ICU discharge.
  Interventions: Other: Passive Range of Motion

INTERVENTIONS:
Other: Early and Active Physical Therapy — Cycle-ergometer exercise will be performed in the more active manner tolerated by patient. Potency attained will be registered during 30 min of exercise.
  Our physiotherapy protocol includes also others exercises like ambulation with assistance, cycle-ergometer for arms and legs, etc.
  Other Names: Early Physical Rehabilitation; Early Physical Training; Early Physiotherapy; Early Mobilization; Very Early Mobilisation; Early Exercise; Early Activity; Early Mobility Therapy
  Arms: Intervention Group
Other: Passive Range of Motion — Passive mobilization will be performed in all limbs as 10 repetitions of every range of motions. Extension position will be maintained for some seconds to attaint muscular elongation in every muscular group.
  Other Names: Passive Range of Motion (PROM); Passive Mobilization; Articular mobilization; Routinary Passive Range of Motion; Usual manual mobilization

SUMMARY:
It is clearly shown that patients in the Intensive care Unit (ICU) with severe sepsis or multi organic failure are very susceptible to develop neuromuscular complications. That can be attributed to a hyper catabolic state, general inflammation and immobilization. This can leads a significant muscle wasting, polyneuropathy and/or myopathy. These alterations have been defined with the term Intensive Care Acquired Weakness (ICUAW) and can leads important functional squeals and impaired quality of life for months, years and in some cases irreversibly.

To overcome these complications, early activation by physiotherapy becomes an important tool. This type of treatment has been show to be feasible, safe and improves the functional capacity of patients. In addition to a reduction in the duration of ICU and hospital stay and improved quality of life for patients.

The objective of this study is to demonstrate that the early and active physical activity in patients with severe sepsis can limit the loss of muscle mass and complications related to this type of damage.

Procedures: Patients or relatives will be asked to participate in the study. If a positive response is done, patients will be randomized in an intervention or control group.

A baseline evaluation will be performed during the first day of study admission. That includes a physical exploration, electrophysiological studies, skeletal muscle histological/biochemical evaluations and monitoring of blood biomarkers and others clinical outcomes will be registered.

Intervention will be divided in a morning and afternoon times, patient will be positioned in chair or bed and mobilized by physiotherapist. As usual, all patients will be attaining manual mobilization for 20 minutes twice a day. Only for intervention group, additional cycle-ergometer exercise will be performed for 30 minutes at better performance achieved and tolerated for patient. All vitals parameters will be strictly controlled before, during and after intervention.

The same baseline evaluation will be repeated after day 7 and clinical outcomes will be registered until ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable patients.
* Admitted to ICU for sepsis or MOF (multiple organ failure) or who developing during their ICU stay within the first 24 hours of the ICU admission.
* With an expected ICU stay of at least 7 days.

Exclusion Criteria:

* Patients without approved consent.
* Patients with a known neuromuscular disorder before ICU admission.
* Moribund patients.
* Severe metabolic/hemodynamic instability despite pharmacological support.
* Having conditions that impair evaluation techniques or intervention methods.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in activation of skeletal muscle synthetic and catabolic pathways. | Within the first 7 days (plus or minus 1 days)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François Laterre, Professor, Study Chair — Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc)
Locations (1):
- Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc), Brussels, Brussels Capital, Belgium

REFERENCES:
- [Derived] Hickmann CE, Castanares-Zapatero D, Deldicque L, Van den Bergh P, Caty G, Robert A, Roeseler J, Francaux M, Laterre PF. Impact of Very Early Physical Therapy During Septic Shock on Skeletal Muscle: A Randomized Controlled Trial. Crit Care Med. 2018 Sep;46(9):1436-1443. doi: 10.1097/CCM.0000000000003263. PMID 29957714